CLINICAL TRIAL: NCT01364688
Title: Randomized Control Trial of Oral Alfacalcidol and Coronary Artery Calcification in Predialysis Chronic Kidney Disease
Brief Title: Oral Alfacalcidol and Coronary Artery Calcification in Predialysis Chronic Kidney Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Sinee Disthabanchong, MD, Division of Nephrology, Department of Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-05-2011
Record Dates: First submitted 2011-05-26; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Vascular Calcification
Keywords: coronary calcification; vascular calcification; active vitamin D; alfacalcidol
MeSH Terms: conditions — Vascular Calcification | interventions — alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): oral alfacalcidol
  Interventions: Drug: oral alfacalcidol
- Control (No Intervention): No drug
  Interventions: Drug: no drug

INTERVENTIONS:
Drug: oral alfacalcidol — Oral alfacalcidol 0.5 microgram per day
  Arms: Treatment
Drug: no drug — no drug
  Arms: Control

SUMMARY:
Active vitamin D at therapeutic dose may prevent vascular calcification but in supraphysiologic dose may precipitate it.

DETAILED DESCRIPTION:
Active vitamin D compound is used frequently in the treatment of hyperparathyroidism in chronic kidney disease. Recent evidence from animal studies suggested that low dose of active vitamin D may be protective against vascular calcification, whereas high dose could precipitate it. The present study will examine the effect of low dose oral alfacalcidol on coronary artery calcification in predialysis chronic kidney disease patients with hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Predialysis chronic kidney disease with GFR < 90 mL/min/1.73m2
* PTH above the upper limit of normal
* serum calcium and phosphate below the upper limit of normal

Exclusion Criteria:

* changes in GFR>15% during the past 3 months
* receive elemental calcium>500 mg/day
* currently taking active vitamin D, oral calcium with elemental calcium>500 mg/day or bisphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in Coronary Artery Calcification | 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Phayathai, Bangkok, Thailand